CLINICAL TRIAL: NCT06277492
Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics of Single and Multiple Ascending Oral Doses of SUL-238 in Healthy Subjects
Brief Title: A First-In-Human Study of Single and Multiple Ascending Doses of Oral SUL-238 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GEN İlaç ve Sağlık Ürünleri A.Ş. (Industry)
Collaborators: Sulfateq B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GN-001
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
Keywords: SUL-238; Oral; Safety; Pharmacokinetics; Food effect
MeSH Terms: interventions — Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Single dose SUL-238 (Active Comparator): PART 1: Single ascending oral doses of SUL-238 (50 mg, 100 mg, 250 mg, 500 mg, 1000 mg and 2000 mg)
  Interventions: Drug: Single ascending doses SUL-238
- Single dose placebo (Placebo Comparator): PART 1: Single oral dose of placebo
  Interventions: Drug: Single dose Placebo
- Single dose pharmacokinetics of SUL-238 (Experimental): PART 2: Single oral dose of SUL-238 (at maximum tolerated dose)
  Interventions: Drug: Single dose SUL-238
- Multiple doses SUL-238 (Active Comparator): PART 3: Multiple ascending oral doses of SUL-238 (at maximum tolerated dose and 1 dose level lower than MTD)
  Interventions: Drug: Multiple ascending doses SUL-238
- Multiple doses placebo (Placebo Comparator): PART 3: Multiple oral doses of placebo
  Interventions: Drug: Multiple doses Placebo
- Single dose pharmacokinetics of SUL-238 (food effect) (Active Comparator): PART 2B: 2000 mg single oral dose of SUL-238
  Interventions: Drug: 2000 mg SUL-238 single dose for pharmacokinetics (food effect)
- Single dose Placebo (food effect) (Placebo Comparator): PART 2B: Single oral dose of placebo
  Interventions: Drug: Single dose placebo (food effect)

INTERVENTIONS:
Drug: Single ascending doses SUL-238 — PART 1: SUL-238 single ascending doses
  Arms: Single dose SUL-238
Drug: Single dose Placebo — PART 1: Placebo single dose
  Arms: Single dose placebo
Drug: Single dose SUL-238 — PART 2: SUL-238 single dose for pharmacokinetics
  Arms: Single dose pharmacokinetics of SUL-238
Drug: Multiple ascending doses SUL-238 — PART 3: SUL-238 multiple ascending doses
  Arms: Multiple doses SUL-238
Drug: Multiple doses Placebo — PART 3: Placebo multiple doses
  Arms: Multiple doses placebo
Drug: 2000 mg SUL-238 single dose for pharmacokinetics (food effect) — PART 2B: 2000 mg single dose of SUL-238
  Arms: Single dose pharmacokinetics of SUL-238 (food effect)
Drug: Single dose placebo (food effect) — PART 2B: Placebo single dose
  Arms: Single dose Placebo (food effect)

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, single-center study is to evaluate the safety, tolerability, pharmacokinetics of single and multiple oral doses of SUL-238 in healthy subjects (aged ≥40 years).

DETAILED DESCRIPTION:
This double-blind placebo-controlled study will be completed in 4 parts.

Part 1 will be single ascending dose in which 6 different oral doses (50 mg, 100 mg, 250 mg, 500 mg, 1000 mg and 2000 mg) will be administered to healthy adult male subjects. Each dosing group, including dose escalations, will be performed as described below:

Dose escalation will be performed until suspected adverse events (AEs) are observed. AEs will be evaluated by the blinded investigator, based on clinical signs detailed in the MedDRA criteria. At each dose level, 2 subjects will be administered SUL-238, whereas 1 subject will be administered the placebo. Escalation to the next higher dose level may occur only if no treatment-emergent AEs are observed in the 2 subjects that received SUL-238. If 1 out of 2 subjects experiences a suspected AE, 5 new subjects will be enrolled at the same dose level (4 subjects will receive one SUL-238 tablet and 1 subject will receive one placebo tablet). If no further suspected AEs occur, escalation to the next higher dose level will be performed. If any additional suspected AE is noted, dose escalation is stopped, and the previous dose level is considered the maximum tolerated dose (MTD). If suspected AE are observed in 2 subjects, dose escalation will be stopped and 5 new subjects (4 subjects will receive one SUL-238 tablet and 1 subject will receive one placebo tablet) will be enrolled at the next lower dose level. If no further suspected AE are observed, this dose level is considered the MTD.

Part 2 of the study will be single dose pharmacokinetics study in which 1 dose level below that with suspected AEs will be administered to 10 healthy adult male or female subjects (aged ≥40 years). Five male subjects and 5 female subjects will receive SUL-238. After obtaining the initial PK results from Part 1, at least 3 volunteers who accept to be tapped for Cerebrospinal Fluid (CSF) collection will provide one CSF sample on Day 1, at the time point of 1 hour after reaching Cmax during Part 2 of the study.

Part 2B will be a randomized, single-dose, two-treatment, two-period, crossover study. A total of twenty (20) healthy adults (10 male and 10 female volunteers, aged ≥40 years) will be included. The volunteers will be randomized equally into two treatment groups (each group will have 5 male and 5 female volunteers) in the first period: fasted versus high-fat-fed. All volunteers will receive a single dose of 2000 mg SUL-238 either in a fasted state (at least 10 hours) or after consuming a standardized high-fat meal (30 minutes before the study drug). In the second period, which will be conducted 14 days after the first period (washout period), a crossover will be implemented: volunteers who received SUL-238 in a fasted state in the first period will receive 2000 mg SUL-238 after a high-fat meal in the second period, and vice versa. A high-fat meal will have a total of 800-1000 calories, with ≥50% (500-600 calories) coming from fat. At least three volunteers in each group who accept to be tapped for CSF collection will provide one CSF sample on Day 1, at the time point of 1 hour after reaching Cmax during Part 2B of the study.

Part 3 of the study will be multiple ascending oral doses of SUL-238 or placebo in which 30 healthy elderly subjects (aged ≥40 years) will be included. There will be 2 dosing groups (n=15 for each) once (or twice, or three times a day) daily (5 male subjects and 5 female subjects) in each dosing group for SUL-238, dosing regimen and doses of SUL-238 will be decided after Part 2B. The volunteers will stay at the investigational site for up to 72 hours following the initial dosing (Day 1-4) as well as after the final dosing (Day 14-17). After completion of 72-hour visit, volunteers will be discharged from the clinical unit. The treatment regimen spans a 14-day period, during which participants will undergo continuous monitoring for an additional 14 days. A daily clinic visit will be required from volunteers for the administration of the investigational medicine until day 14. The MTD will be the dose for the first dosing group. The second dosing group will be one below the MTD level (e.g., if MTD is 2000 mg, the second dosing group will receive 1000 mg SUL-238). In the first dosing group three 3 male and 2 female subjects and in the second dosing group 2 male and 3 female subjects will receive placebo. PK parameters as well as renal clearance and percentage of drug excreted in urine and feces will be measured in both dosing groups. At least 3 volunteers who agreed to be tapped for a CSF in both dosing groups receiving SUL-238 will provide one CSF sample on day 14 (post-first dose) 8 or 12 hours post-morning dose in Part 3.

In Part 1, 2 and 2B blood samples will be drawn, before drug administration (0 hours), after 30 minutes and at the following time points: 1, 2, 4, 8, 12, 18, 24, 32, 48 and 72 hours. In Part 3, blood samples will be drawn, before drug administration (0 hours), after 30 minutes and at the following time points: 1, 2, 4, 6, 8, 12, 18, 24, 32, 48 and 72 hours, Days 8 (pre-morning dose), 14 (pre-last dose baseline, post-last dose at 30 minutes, 1, 2, 4, 6, 8, 12 and 18 hours), 15 (post-last dose at 24 and 32 hours), 16 and 17. The subject randomized to placebo arm will provide blood samples as subjects randomized to active drug.

In Part 1 and 2 ambulatory visits will be performed at Day 8, 11, 15, 22 and 29 after dosing on which volunteers will visit the clinical investigational site. In Part 2B ambulatory visits will be performed at Day 8, 22 and 29 after dosing. The volunteers will be followed up until Day 29. In Part 3, ambulatory visits will be performed at Day 22, and 29 after dosing on which volunteers will visit the clinical investigational site.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests and cardiac monitoring.
2. Men and women aged≥40 years at Screening.
3. Subject must understand the nature of the study and provide signed and dated written informed consent in accordance with local regulations before the conduct of any study-related procedures.
4. Able to complete all study related testing and evaluations.
5. Women and men of child-bearing potential with partners of child-bearing potential must agree to use highly effective contraception. For male subjects, contraception should continue for 90 days after the last dose of investigational medicinal product (IMP, one spermatic cycle).
6. Women of non-childbearing potential must be post-menopausal (the last menstrual period was at least 12 months ago, and follicle-stimulating hormone [FSH] at Screening confirms post-menopausal status), or have no uterus, ovaries, or fallopian tubes (or have their fallopian tubes tied). All women must have a negative pregnancy test result before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
7. Body weight > 50 kg for men and > 50 kg for women and Body Mass Index (BMI) within the range 18.5-30.0 kg/m2, inclusive.
8. Subject must be, in the opinion of the Investigator, able to participate in all scheduled evaluations, likely to complete all required tests, and likely to be compliant.

Exclusion Criteria:

1. A positive urine drug screen/alcohol breath test at Screening or Day -1.
2. Any history of intellectual disability or psychiatric disorders, including substance use disorders, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, except a history of mild depression/anxiety that has been resolved for at least the past 12 months.
3. A positive Hepatitis B surface antigen, Hepatitis C antibody, or Human Immunodeficiency Virus (HIV) antibody test at Screening.
4. Alanine aminotransferase or aspartate aminotransferase levels greater than 1.5 times the upper limit of normal (ULN) at Screening or between Screening and first dose administration.
5. History of regular alcohol consumption within the last 12 months, defined as an average weekly intake of >21 alcoholic drinks/week for men or >14 alcoholic drinks/week for women.
6. Regularly consumed (e.g., more days than not) excessive quantities of xanthine-containing beverages (e.g., more than five cups of coffee or the equivalent per day) within 30 days prior to Day -1.
7. Received or used an investigational product (including placebo) or device within the following time period prior to Day -1 in the current study: 90 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
8. Use of prescription or non-prescription drugs, vitamins, herbal, and dietary supplements within 7 days (or 28 days if the drug is a potential hepatic enzyme inducer) or 5 half-lives (whichever is longer) prior to Day -1.
9. History of clinically significant sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
10. A positive serum pregnancy test or lactation.
11. A history or presence of any disease, condition, or surgery likely to affect drug absorption, distribution, metabolism, or excretion. Subjects with a history of cholecystectomy should be excluded.
12. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, pulmonary, ophthalmologic, immunologic, hematologic, dermatologic, or neurologic abnormality.
13. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgement of the Investigator or Medical Monitor, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
14. A clinically significant vital signs abnormality at Screening or Day -1 This includes, but is not limited to, the following, in the sitting position (3 measurements, each 5 minutes apart): (a) systolic blood pressure < 90 or >140 mmHg, (b) diastolic blood pressure < 50 or > 95 mmHg, or (c) heart rate < 45 or > 100 beats per minute.
15. Subjects who have previously been enrolled in this study.
16. The subject is, in the opinion of the Investigator or Medical Monitor, unlikely to comply with the protocol or is unsuitable for any reason, e.g., known issues with ability to swallow tablets.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as Measured by NCI-CTCAE criteria | Up to day 29
  The safety and tolerability of SUL-238 will be assessed by documenting adverse events occurring after single dose administration on Day 1 in Part 1, Part 2 and Part 2B until Day 29. After once daily continuous dosing of SUL-238 for 14 Days in Part 3, the safety and tolerability of SUL-238 will be assessed by documenting adverse events occurring after during multiple dose administrations until Day 29. There will be no dosing between Day 15 and 29 in Part 3.
Incidence of Treatment-Emergent Adverse Events as Measured by Clinical Laboratory Measurements According to Established Clinical Normal Ranges | Up to day 29
  Clinical laboratory tests include hematology and clinical chemistry including renal function tests, hepatic enzymes, electrolytes and creatine kinase.
  * Change from baseline (pre-dose sample) at 24 hours (Day 2) and Days 3, 4, 8, 15 and 29 post-dose of SUL-238 (Part 1, Part 2).
  * Change from baseline (pre-dose sample) at 24 hours (Day 2) and Days 3, 4, 8, and from Day 14 (pre-second dose baseline), at 24 hours post-second dose (Day 16), and Days 17, 18, 22 and 29 post-first dose of SUL-238 (Part 2B).
  * Change from baseline (pre-dose sample) at 24 hours (Day 2) and at Days 3, 4, 8, 14 (1 hour post-last dose), 15 (24 hours post-last dose), 16, 17, 22 and 29 post-first dose SUL-238 for Part 3.
  * Blood and urine samples will be taken after administration of SUL-238 and values will be compared to baseline and established normal ranges to determine how SUL-238 administration impacts normal body function.
Incidence of Treatment-Emergent Adverse Events as Measured by ECG | Up to day 29
  * As compared to baseline (an ECG taken at 60 minutes pre-dose); ECG evaluations will be performed at 30 minutes, 1 hour, 12 hours post-dose and Days 2 (24 hours), 3, 4, 8, 15 and 29 post-dose of SUL-238 occurring after single dose administration (Part 1 and Part 2).
  * As compared to baseline (an ECG taken at 60 minutes pre-dose); ECG evaluations will be performed at 30 minutes, 1 hour, 12 hours post-first dose and Days 2 (24 hours), 3, 4, as well as Days 15 (at 60 minutes pre-second dose and at 30 minutes, 1 hour, 12 hours post-second dose), 16 (24 hours post-second dose), 17, 18, 22, and 29 (Part 2B).
  * As compared to baseline (an ECG taken at 60 minutes pre-dose); ECG evaluations will be performed at 30 minutes, 1 hour, 12 hours post-dose and Days 2 (24 hours), 3, 4, 8, 14 (1-hour post-last dose), 15, 16, 17, 22, and 29 post-dose SUL-238 for Part 3.
Incidence of Treatment-Emergent Adverse Events as Measured by physical examination and vital signs | Up to day 29
  Vital signs include blood pressure, heart rate and oral temperature. Change from baseline at every time points defined for Part 1, Part 2, Part 2B, and Part 3 until Day 29 post-first dose of SUL-238.
Incidence of Treatment-Emergent Adverse Events as Measured by central nervous system (CNS) and autonomic nervous system (ANS) examination. | Up to day 29
  After each dose of SUL-238 through completion of dosing, up to Day 29 in Part 1, Part 2, Part 2B, and Part 3, at all timepoints defined for the evaluation of adverse events, CNS and ANS examinations will be performed, and outcomes will be documented. CNS examinations should include evaluation of mental status, cranial and peripheral nerves, muscle strength, gait and coordination, sensations and reflexes. For the evaluation of ANS, the presence of postural hypotension, heart rate changes, pupil reflex change to light and signs and symptoms of decreased or absent sweating should be checked.

SECONDARY OUTCOMES:
PK parameter: Maximum drug concentration in plasma (Cmax) of SUL-238 after a single ascending dose (Part 1 and Part 2). | Part 1 and Part 2: Up to day 4
  Blood collection on Days 1, 2, 3 and 4. On Day 1 (pre-dose baseline, post-dose at 30 minutes, 1, 2, 4, 8, 12 and 18 hours), and Days 2 (24 and 32 hours post-dose), 3 (48 hours post-dose), and 4 (72 hours post-dose).
Food effect on PK parameter: Maximum drug concentration in plasma (Cmax) of SUL-238 after a single dose (Part 2B). | Up to day 18
  Blood collection on Days 1, 2, 3, 4, 15, 16, 17, and 18. On Day 1 (pre-dose baseline, post-dose at 30 minutes, 1, 2, 4, 8, 12 and 18 hours), and Days 2 (24 and 32 hours post-dose), 3 (48 hours post-dose), 4 (72 hours post-dose), and after cross-over on second period on Days 15 (pre-second dose baseline, post-second dose at 30 minutes, 1, 2, 4, 8, 12 and 18 hours), 16 (24 and 32 hours post-second dose), 17 (48 hours post-second dose), and 18 (72 hours post-second dose).
PK parameter: Maximum drug concentration in plasma (Cmax) of SUL-238 after multiple ascending doses (Part 3). | Part 3: Up to day 17
  Blood collection on Days 1, 2, 3, 4, 8, 14 (pre-last dose), 15, 16 and 17. On Day 1 (pre-first dose baseline, post-first dose at 30 minutes, 1, 2, 4, 6, 8, 12 and 18 hours), Days 2 (24 and 32 hours post-first dose), 3 (48 hours post-first dose), 4 (72 hours post-first dose), 8, 14 (pre-last dose baseline, post-last dose at 30 minutes, 1, 2, 4, 6, 8, 12 and 18 hours), 15 (24 and 32 hours post-last dose), 16 (48 hours post-last dose), and 17 (72 hours post-last dose).
PK parameter: Area under the concentration-time curve in plasma (AUC) of SUL-238 after single ascending dose (Part 1 and Part 2). | Part 1 and Part 2: Up to day 4
  Blood collection on Days 1, 2, 3 and 4. On Day 1 (pre-dose baseline, post-dose at 30 minutes, 1, 2, 4, 8, 12 and 18 hours), Days 2 (24 and 32 hours post-dose), 3 (48 hours post-dose), and 4 (72 hours post-first dose). The determination of the Area under the concentration-time curve will be made from the data of pre-dose (time 0) to the time of the last quantifiable concentration (tlast) and from pre-dose (time 0) extrapolated to infinite time (AUClast + Clast/λz) calculated using the linear-log trapezoidal rule.
Food effect on PK parameter: Area under the concentration-time curve in plasma (AUC) of SUL-238 after single dose in each period (Part 2B). | Up to day 18
  Blood collection on Days 1, 2, 3, 4, 15, 16, 17, and 18. On Day 1 (pre-dose baseline, post-dose at 30 minutes, 1, 2, 4, 8, 12 and 18 hours), Days 2 (24 and 32 hours post-dose), 3 (48 hours post-dose), and 4 (72 hours post-first dose). On Day 15 (pre-second dose baseline, post-second dose at 30 minutes, 1, 2, 4, 8, 12 and 18 hours) and Days 16 (24 and 32 hours post-second dose), 17 (48 hours post-second dose), and 18 (72 hours post-second dose). The determination of the Area under the concentration-time curve will be made from the data of pre-dose (time 0) to the time of the last quantifiable concentration (tlast) and from pre-dose (time 0) extrapolated to infinite time (AUClast + Clast/λz) calculated using the linear-log trapezoidal rule (for each period data).
PK parameter: Area under the concentration-time curve in plasma (AUC) of SUL-238 after multiple ascending doses (Part 3). | Part 3: Up to day 17
  Blood collection on Days 1, 2, 3, 4, 8, 14 (pre-last dose), 15, 16, and 17. On Day 1 (pre-first dose baseline, post-first dose at 30 minutes, 1, 2, 4, 6, 8, 12 and 18 hours), Days 2 (24 and 32 hours post-first dose), 3 (48 hours post-first dose), 4 (72 hours post-first dose), 8, 14 (pre-last dose baseline, post-last dose at 30 minutes, 1, 2, 4, 6, 8, 12 and 18 hours), 15 (24 and 32 hours post-last dose), 16 (48 hours post-last dose), and 17 (72 hours post-last dose). The determination of the area under the concentration-time curve will be made from the data of pre-dose (time 0) to the time of the last quantifiable concentration (tlast) and from pre-dose (time 0) extrapolated to infinite time (AUClast + Clast/λz) calculated using the linear-log trapezoidal rule.
Renal clearance and percentage of drug excreted in urine after single and multiple ascending doses of SUL-238. | Part 1 and Part 2: Up to day 2, Part 2B: Up to day 16 and Part 3: Up to day 15
  Part 1 and 2: On Day 1 (pre-dose baseline), and 0-4, 4-8, 8-12, 12-24 hours and on Day 2 (24-48 hours) in 24 hours urine samples post-dose.
  Part 2B: On Day 1 (pre-dose baseline), and 0-4, 4-8, 8-12, 12-24 hours and on Day 2 (24-48 hours) in 24 hours urine samples post-dose. On Day 15 (pre-second dose baseline), and 0-4, 4-8, 8-12, 12-24 hours and on Day 16 (24-48 hours) in 24 hours urine samples post-second dose.
  Part 3: On Day 1, (pre-dose baseline), and 0-4, 4-8, 8-12, 12-24 hours and post-first dose on Day 2 (24-48 hours) in 24 hours urine samples, Day 8 (24 hour sample), 14 (pre-last dose baseline), and 0-4, 4-8, 8-12, 12-24 hours (post-last dose), 15 (24-48 hours) (post-last dose in 24 hours urine samples). The determination of the renal clearance and amount of SUL-238 excreted in urine will be measured.
Percentage of drug excreted in feces after multiple ascending doses of SUL-238. | Part 3: Up to day 29
  Part 3: Baseline (pre-first dose), Days 2 (24 hours post first-dose), 8, 15 (24 hours post last-dose), 22, and 29. The amount of SUL-238 excreted in feces will be determined.
The cerebrospinal fluid (CSF) levels of SUL-238 | Part 2 and Part 2B: Day 1 and Part 3: Day 8
  Based on the time to reach Cmax value obtained in Part 1, the cerebrospinal fluid (CSF) levels of the investigational drug will be evaluated through collection of CSF samples and evaluation of SUL-238 concentrations during Part 2, Part 2B and Part 3 of the study. The CSF collections will be performed on Day 1 (dosing day) in Part 2 and Part 2B at a time point which will be defined as one hour after the time point when the Cmax is reached (Tmax) and on Day 14 (post-first dose) at 8 or 12 hours post-morning dose in Part 3. Due to its invasive nature, this evaluation will only be performed based on the acceptance of the healthy volunteers and CSF samples will be collected from the volunteers receiving SUL-238.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Sezer, MD, Principal Investigator — Department of Pharmacology, Faculty of Medicine, Erciyes University
Locations (1):
- Erciyes University IKUM Center, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No